CLINICAL TRIAL: NCT03561987
Title: Identification of Biomarkers Derived From Adipose Tissue With Potential Utility in the Diagnosis and Prognosis of Cardiovascular Risk of the Obese Patient.
Brief Title: Biomarkers Derived From Adipose Tissue Useful for Diagnosis and Prognosis of Cardiovascular Risk (CVR) in Obese Patient
Acronym: CROP
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado (Other Government)
Responsible Party: Principal Investigator, Juan Antonio Suárez Cuenca, Ph.D. in Biomedical sciences, Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado
Other Study IDs: 386.2013
Record Dates: First submitted 2018-06-08; First posted 2018-06-19 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-06

CONDITIONS: Metabolic Syndrome; Diabetes Mellitus; Inflammatory Response
Keywords: ADIPOSE TISSUE, CARDIOVASCULAR, OBESE PATIENTS
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Biospecimen Retention: Samples With DNA — Subcutaneous adipose tissue, visceral adipose tissue, liver tissue, blood samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Obese patients and bariatric surgery: The investigators include men and women, over 18 years old, with morbid obesity and candidates for bariatric surgery, under the routine of the treating service, with signature of acceptance of your participation, by informed consent.
  The investigators exclude patients with medication with potential effect on adipose tissue or cardiovascular risk in the last month, also with severe infections in the last month or clinically unstable conditions.
  Patients are eliminated in the study if they dont have the desire to continue in the study, and if the samples or the information are insufficient for an adequate analysis.
  Interventions: Procedure: Bariatric surgery
- No obese patients and abdominal surgery: The investigators include men and women, over 18 years old, without obesity and candidates for abdominal surgery (hernioplasty, cholecystectomy, fundoplication), under the routine of the treating service, with signature of acceptance of your participation, by informed consent.
  The investigators exclude patients with medication with potential effect on adipose tissue or cardiovascular risk in the last month, also with severe infections in the last month or clinically unstable conditions.
  Patients are eliminated in the study if they dont have the desire to continue in the study, and if the samples or the information are insufficient for an adequate analysis.
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — There are two components to the procedure. First, a small stomach pouch, approximately one ounce or 30 milliliters in volume, is created by dividing the top of the stomach from the rest of the stomach. Next, the first portion of the small intestine is divided, and the bottom end of the divided small intestine is brought up and connected to the newly created small stomach pouch. The procedure is completed by connecting the top portion of the divided small intestine to the small intestine further down so that the stomach acids and digestive enzymes from the bypassed stomach and first portion of small intestine will eventually mix with the food.

SUMMARY:
This study evaluates the relationship between the adipose tissue, as an active component, which can define metabolic phenotypes linked to cardiovascular risk modification post bariatric surgery.

DETAILED DESCRIPTION:
Bariatric surgery induces a significant reduction in co-morbidities associated with obesity, such as Diabetes mellitus, dyslipidemia, liver disease, arterial hypertension, obstructive apnea and cardiovascular risk. However this does not happen in all obese patients, even when there is a weight reduction.

It is known that the adipose tissue is actively involved in synthesis of cytokines and its role in metabolic phenotypes has been suggested. It is possible that the intrinsic mechanisms of adipose tissue participate in several benefits observed in morbidly obese patients who undergo to an anti-obesity surgery.

So this study explores the involvement of adipose tissue as an active component, which can define metabolic phenotypes linked to cardiovascular risk modification post bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old.
* Morbid obese patients candidates to bariatric surgery.

Exclusion Criteria:

* Second bariatric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Morbid obese patients candidates to bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2013-11-06 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2022-01-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate the association of the cardiovascular benefit of the obese patient after bariatric surgery with the basic mechanisms of adipose tissue (metabolic profile) | 3 years
  Evaluate the association of the cardiovascular benefit of the obese patient after bariatric surgery with the basic mechanisms of adipose tissue (metabolic profile)

SECONDARY OUTCOMES:
Correlation between serum concentration of pro-inflammatory biomarker and the reduction of subclinical endothelial disfunction. | 9 months
  measurements of carotid intima-media thickness (CIMT) in millimeter and Flow mediated dilatation (FMD) in percent in a basal time and see over time the reduction (if any) of those endothelial markers
Determine the association of the cardiovascular prognosis modification (risk subgroups) with the basal metabolic profile. | 9 months
  After the 9 months follow up, the authors will correlated the pro-inflammatory cytokines, presence or absence of adipose proteins.

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT03561987/Prot_SAP_000.pdf